CLINICAL TRIAL: NCT01752907
Title: Randomized, Single-blind Study to Estimate the Effect of Patient Education on Reported Bone Pain in Breast Cancer Patients Receiving Chemotherapy and Pegfilgrastim
Brief Title: Effect of Patient Education on Reported Bone Pain in Breast Cancer Patients Receiving Chemotherapy and Pegfilgrastim
Acronym: VINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20110148
Record Dates: First submitted 2012-11-15; First posted 2012-12-19 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chemotherapy; Pegfilgrastim; Neulasta; Bone Pain; Education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Education DVD (Experimental): Participants received chemotherapy and pegfilgrastim administered as a single subcutaneous injection dose of 6 mg 24 to 72 hours after chemotherapy. Participants were required to watch a general chemotherapy side effects education DVD on 2 separate visits to the clinic prior to the first administration of pegfilgrastim in cycle 1.
  Interventions: Other: General Education DVD
- Bone Pain Education DVD (Experimental): Participants received chemotherapy and pegfilgrastim administered as a single subcutaneous injection dose of 6 mg 24 to 72 hours after chemotherapy. Participants were required to watch a bone pain education DVD on 2 separate visits to the clinic prior to the first administration of pegfilgrastim in cycle 1.
  Interventions: Other: Bone Pain Education DVD

INTERVENTIONS:
Other: General Education DVD — A general chemotherapy side effects education DVD
  Arms: General Education DVD
Other: Bone Pain Education DVD
  Arms: Bone Pain Education DVD

SUMMARY:
The purpose of this study is to determine if patient education can affect patient reported bone pain in breast cancer patients receiving chemotherapy and pegfilgrastim.

DETAILED DESCRIPTION:
In this study, the effect of patient education on reported bone pain in breast cancer patients receiving adjuvant or neoadjuvant chemotherapy and pegfilgrastim will be investigated.

Each patient will receive adjuvant or neoadjuvant chemotherapy with pegfilgrastim prophylaxis, beginning in the first cycle and continuing throughout the study period. The study period for this study is the first 4 cycles of chemotherapy. participants can be planning to receive regimens with > 4 cycles, but data will only be collected for the first 4 cycles. The choice of chemotherapy regimen (agent, dose, and schedule) is at the discretion of the treating physician. Commercially available pegfilgrastim will be administered according to US Prescribing Information and is considered background therapy.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or over
* Eastern cooperative oncology group (ECOG) performance status 0-2
* Female with newly diagnosed, not previously treated with chemotherapy, stage I-III breast cancer
* Planning to receive at least 4 cycles of adjuvant or neoadjuvant chemotherapy
* Medically eligible to safely receive adjuvant or neoadjuvant chemotherapy and pegfilgrastim as determined by the investigator
* Planning to receive prophylaxis with pegfilgrastim starting in the first cycle and continuing throughout each chemotherapy cycle of the study period
* Has provided informed consent
* Able to understand the content of the DVD material, in investigator's opinion
* Able to read and understand English

Exclusion Criteria

* Planning to receive weekly chemotherapy
* Chronic use of oral non-steroidal anti-inflammatory drugs (NSAIDs) or oral antihistamines with the following exception:

  - Chronic oral aspirin use for cardiovascular-related indications
* Ongoing chronic pain, or other painful conditions requiring treatment (including immediate post-operative treatment of surgical or procedural-associated pain) as determined by the investigator
* Chronic oral steroid use. Premedication related to the administration of taxanes, and use of anti-emetics is allowed, per usual clinical practice.
* Prior chemotherapy treatment for cancer within 5 years of current breast cancer diagnosis
* Prior use of granulocyte-colony stimulating factor (G-CSF)
* Currently enrolled in, or less than 30 days since ending, another clinical trial which includes language directing G-CSF (filgrastim, pegfilgrastim, other) or granulocyte-macrophage colony stimulating factor (GM-CSF) (sargramostim) use
* Currently enrolled in, or less than 30 days since ending, another interventional clinical trial which includes a blinded treatment or blinded treatment arm (whether or not the subject is randomized to the blinded arm)
* Currently enrolled in, or less than 30 days since ending, another interventional clinical trial which includes the use of any agent not currently considered to be standard therapy for the adjuvant or neoadjuvant treatment of stage I-III breast cancer based on National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Breast Cancer
* Currently enrolled in, or less than 30 days since ending, any pain intervention study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2014-12-15 (Actual); Study Completion 2014-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (51):
- United States (51):
  - Research Site, Fountain Valley, California
  - Research Site, Mission Hills, California
  - Research Site, Santa Rosa, California
  - Research Site, Vallejo, California
  - Research Site, Whittier, California
  - Research Site, Danbury, Connecticut
  - Research Site, Greenwich, Connecticut
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Mason City, Iowa
  - Research Site, Mount Sterling, Kentucky
  - Research Site, Lewiston, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Fairhaven, Massachusetts
  - Research Site, Lansing, Michigan
  - Research Site, Robbinsdale, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Jefferson City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Englewood, New Jersey
  - Research Site, Hamilton, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Vineland, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Cooperstown, New York
  - Research Site, Glens Falls, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Suffern, New York
  - Research Site, Asheboro, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Goldsboro, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Bend, Oregon
  - Research Site, Gettysburg, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Aberdeen, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, El Paso, Texas
  - Research Site, Danville, Virginia
  - Research Site, Burien, Washington

REFERENCES:
- [Background] Guinigundo AS, Maxwell CL, Vanni L, Morrow PK, Reiner M, Shih A, Klippel Z, Blanchard E. A Randomized, Single-Blind Study Evaluating the Effect of a Bone Pain Education Video on Reported Bone Pain in Patients with Breast Cancer Receiving Chemotherapy and Pegfilgrastim. Pain Manag Nurs. 2018 Dec;19(6):693-706. doi: 10.1016/j.pmn.2018.04.002. Epub 2018 Jun 21. PMID 29935909
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 48 centers in the United States. Patients with stage I to III breast cancer planning to receive standard neoadjuvant or adjuvant chemotherapy regimens with pegfilgrastim support for at least 4 cycles were included. The first participant enrolled on 17 January 2013 and the last participant enrolled on 04 September 2014.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive 1 of 2 educational DVDs: general chemotherapy side effects education DVD (GE-DVD) or bone pain education DVD (BP-DVD). Participants remained on study for the first 4 chemotherapy cycles. End of study occurred 30 days after administration of pegfilgrastim in the fourth cycle of chemotherapy.
Period: Overall Study
Arm/Group | General Education DVD | Bone Pain Education DVD
Started | 151 | 153
Received Pegfilgrastim | 149 | 151
Completed | 139 | 133
Not Completed | 12 | 20
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Lost to Follow-up | 2 | 1
Not completed — Decision by Sponsor | 6 | 9

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received primary prophylaxis (cycle 1 administration) with pegfilgrastim.
Groups:
- Total: Total of all reporting groups
Arm/Group | General Education DVD | Bone Pain Education DVD | Total
Number analyzed (Participants) | 149 | 151 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.4) | 54.5 (10.4) | 54.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 151 | 300
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 5 | 6
  Black (or African American) | 19 | 19 | 38
  White | 128 | 124 | 252
  Other | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Patient-reported Bone Pain in Cycle 1
Description: Participants completed a brief bone pain survey once per day for 5 days beginning the day they received their pegfilgrastim injection. The bone pain survey collected the severity of pain using a 0 to 10 scale, where 0 = no pain and 10 indicates worst pain.
Time Frame: Days 1 to 5 during cycle 1.
Population: Full analysis set with imputation
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
units on a scale | 3.2 (0.2) | 3.5 (0.3)
Statistical Analysis 1: Comparison: General Education DVD vs Bone Pain Education DVD; There was no statistical hypothesis testing for this study. The clinical hypothesis was that a difference in mean maximum pain of 0.5 (scale 0 to 10) in favor of bone pain education would be a clinically relevant difference; Test type: Superiority or Other; p = 0.3479, t-test, 2 sided; Treatment Difference = 0.3, 95% CI 2-sided [-0.4 to 1.0], Standard Error of Mean 0.4 — Treatment difference = bone pain DVD - general education DVD

2. Secondary Outcome: Maximum Patient-reported Bone Pain by Cycle and Across All Cycles
Description: as for outcome 1
Time Frame: Days 1-5 for each treatment cycle
Population: Full analysis set with imputation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
units on a scale
  Cycle 2 (n=145, 144) | 2.5 (0.2) | 2.7 (0.3)
  Cycle 3 (n=142, 139) | 2.7 (0.2) | 2.6 (0.2)
  Cycle 4 (n=141, 133) | 2.4 (0.2) | 2.5 (0.3)
  All Cycles (n-149, 151) | 4.1 (0.3) | 4.6 (0.3)

3. Secondary Outcome: Mean Patient-reported Bone Pain by Cycle and Across All Cycles
Description: as for outcome 1
Time Frame: Days 1-5 for 4 treatment cycles
Population: Full analysis set with imputation
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
units on a scale
  Cycle 1 (n=149, 151) | 1.6 (0.2) | 1.8 (0.2)
  Cycle 2 (n=145, 144) | 1.3 (0.1) | 1.5 (0.2)
  Cycle 3 (n=142, 139) | 1.4 (0.2) | 1.4 (0.2)
  Cycle 4 (n=141, 133) | 1.3 (0.1) | 1.5 (0.2)
  All cycles (n=149, 151) | 1.5 (0.1) | 1.6 (0.1)

4. Secondary Outcome: Patient-reported Bone Pain Area Under the Curve (AUC) by Cycle and Across All Cycles
Description: Patient-reported bone pain AUC was calculated using the trapezoidal rule with bone pain scores from Day 1-5 for each cycle. AUC may range from 0 to 40 per cycle.
Time Frame: Days 1-5 for 4 treatment cycles
Population: Full analysis set with imputation
Measure: Mean (Standard Error); unit: units on a scale * days
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
units on a scale * days
  Cycle 1 (n=149, 151) | 6.7 (0.6) | 7.6 (0.7)
  Cycle 2 (n=145, 144) | 5.4 (0.6) | 6.3 (0.7)
  Cycle 3 (n=142, 139) | 6.2 (0.6) | 6.1 (0.7)
  Cycle 4 (n=141, 133) | 5.6 (0.6) | 6.2 (0.7)
  All Cycles (n=149, 151) | 6.3 (0.6) | 6.6 (0.6)

5. Secondary Outcome: Percentage of Participants With Any Grade Bone Pain as Captured in Standard Adverse Event Reporting
Description: Participants with any grade of bone pain as captured during standard adverse event (AE) reporting. A pre-defined list of Medical Dictionary for Regulatory Activities (MedDRA) version 17.1 preferred terms was used to determine if a participant experienced bone pain: Arthralgia, Arthritis, Back pain, Bone pain, Chest discomfort, Groin discomfort, Limb discomfort, Musculoskeletal chest pain, Musculoskeletal discomfort, Musculoskeletal pain, Neck pain, Non-cardiac chest pain, Osteochondritis Pain, Pain in extremity, Pain in jaw, Pelvic pain, Pubic pain, Sacroiliitis, Spinal pain, Spondylitis.
Time Frame: From randomization until 30 days after the last dose of pegfilgrastim, up to approximately 20 weeks
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
percentage of participants
  Cycle 1 (n=149, 151) | 43.0 | 40.4
  Cycle 2 (n=145, 144) | 37.2 | 35.4
  Cycle 3 (n=142, 139) | 37.3 | 35.3
  Cycle 4 (n= 141, 133) | 38.3 | 37.6
  All cycles (n=149, 151) | 58.4 | 56.3

6. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Bone Pain Captured in Standard Adverse Event Reporting
Description: Participants with grade 3 or 4 bone pain as captured during standard adverse event reporting. A pre-defined list of Medical Dictionary for Regulatory Activities (MedDRA) version 17.1 preferred terms was used to determine if a participant experienced bone pain: Arthralgia, Arthritis, Back pain, Bone pain, Chest discomfort, Groin discomfort, Limb discomfort, Musculoskeletal chest pain, Musculoskeletal discomfort, Musculoskeletal pain, Neck pain, Non-cardiac chest pain, Osteochondritis Pain, Pain in extremity, Pain in jaw, Pelvic pain, Pubic pain, Sacroiliitis, Spinal pain, Spondylitis. The severity of each AE was graded using the Common Terminology criteria for Adverse Events (CTCAE) version 3 and are based on the following:
  Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
Time Frame: From randomization until 30 days after the last dose of pegfilgrastim, up to approximatley 20 weeks.
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
percentage of participants
  Cycle 1 (n=149, 151) | 2.0 | 5.3
  Cycle 2 (n=145, 144) | 0.0 | 2.1
  Cycle 3 (n=142, 139) | 0.0 | 2.2
  Cycle 4 (n=141, 133) | 2.8 | 3.8
  All cycles (n=149, 151) | 4.7 | 6.6

7. Secondary Outcome: Percentage of Participants Who Used Analgesics for the Treatment of Bone Pain by Cycle and Across Cycles
Description: Analgesic use includes both analgesic and non-steroidal anti-inflammatory drugs.
Time Frame: From Day 1 of Cycle 2 until 30 days after the last dose of pegfilgrastim, up to approximately 16 weeks.
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | General Education DVD | Bone Pain Education DVD
Number analyzed (Participants) | 149 | 151
percentage of participants
  Cycle 1 (n=149, 151) | 74.5 | 73.5
  Cycle 2 (n=145, 144) | 69.0 | 65.3
  Cycle 3 (n=142, 139) | 65.5 | 66.2
  Cycle 4 (n=141, 143) | 68.8 | 69.2
  All cycles (n=149, 151) | 85.2 | 80.1

ADVERSE EVENTS:
Time Frame: From randomization until 30 days after the last dose of pegfilgrastim, up to approximately 20 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  All sparticipants included in the analysis received at least one dose of pegfilgrastim.
Groups:
- General Chemotherapy Education DVD: Participants received chemotherapy and pegfilgrastim administered as a single subcutaneous injection dose of 6 mg 24 to 72 hours after chemotherapy. Participants were required to watch a general chemotherapy side effects education DVD on 2 separate visits to the clinic prior to the first administration of pegfilgrastim in cycle 1.
Arm/Group | General Chemotherapy Education DVD | Bone Pain Education DVD
Serious Adverse Events (participants affected / at risk) | 16/149 | 20/151
Other Adverse Events (participants affected / at risk) | 138/149 | 144/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | General Chemotherapy Education DVD (N=149) | Bone Pain Education DVD (N=151)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Localised infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | General Chemotherapy Education DVD (N=149) | Bone Pain Education DVD (N=151)
Anaemia (Blood and lymphatic system disorders) | 23 | 29
Leukocytosis (Blood and lymphatic system disorders) | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 18 | 20
Palpitations (Cardiac disorders) | 2 | 8
Lacrimation increased (Eye disorders) | 8 | 3
Constipation (Gastrointestinal disorders) | 43 | 54
Diarrhoea (Gastrointestinal disorders) | 52 | 51
Dyspepsia (Gastrointestinal disorders) | 14 | 20
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 8
Nausea (Gastrointestinal disorders) | 87 | 86
Oral pain (Gastrointestinal disorders) | 6 | 9
Stomatitis (Gastrointestinal disorders) | 18 | 22
Vomiting (Gastrointestinal disorders) | 21 | 17
Asthenia (General disorders) | 10 | 8
Fatigue (General disorders) | 87 | 97
Mucosal inflammation (General disorders) | 8 | 13
Oedema peripheral (General disorders) | 9 | 14
Pain (General disorders) | 10 | 8
Pyrexia (General disorders) | 12 | 16
Cellulitis (Infections and infestations) | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 8
Urinary tract infection (Infections and infestations) | 7 | 8
Decreased appetite (Metabolism and nutrition disorders) | 28 | 22
Dehydration (Metabolism and nutrition disorders) | 13 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 22
Bone pain (Musculoskeletal and connective tissue disorders) | 47 | 48
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 10
Dizziness (Nervous system disorders) | 11 | 13
Dysgeusia (Nervous system disorders) | 28 | 26
Headache (Nervous system disorders) | 39 | 45
Neuropathy peripheral (Nervous system disorders) | 17 | 11
Anxiety (Psychiatric disorders) | 6 | 15
Insomnia (Psychiatric disorders) | 21 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 49 | 59
Rash (Skin and subcutaneous tissue disorders) | 13 | 10
Flushing (Vascular disorders) | 8 | 5
Hot flush (Vascular disorders) | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.